CLINICAL TRIAL: NCT00919490
Title: A Double-blind, Randomized, Placebo-controlled Phase 1 Study in Healthy Male Adults to Evaluate the Safety, Tolerability and Pharmacokinetic Profiles of Single Dose of ABT-333
Brief Title: A Study of Single Dose of ABT-333 in Healthy Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry)
Responsible Party: Kazuhiko Sawa, Abbott Japan Co., Ltd.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M11-023
Record Dates: First submitted 2009-05-28; First posted 2009-06-12 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-09

CONDITIONS: HCV Infections
Keywords: Healthy Volunteers
MeSH Terms: interventions — dasabuvir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Group 1 (Experimental): Single dose of 400 mg
  Interventions: Drug: ABT-333
- Group 2 (Experimental): Single dose of 800 mg after safety evolution of Group I
  Interventions: Drug: ABT-333
- Group 3 (Experimental): Single dose of 1200 mg after safety evolution of Group 2
  Interventions: Drug: ABT-333
- Group 4 (Experimental): Single dose of 1600 mg after safety evolution of Group 3
  Interventions: Drug: ABT-333
- Group 5 (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-333 — Tablet, see arms for interventional description
  Arms: Group 1; Group 2; Group 3; Group 4
Drug: Placebo — Tablet, see arms for interventional description.
  Arms: Group 5

SUMMARY:
The objectives of this study is to assess the safety, tolerability, and pharmacokinetics of blind, escalating, single, oral doses of ABT-333 under nonfasting conditions in healthy male adult in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent.
* Subject is in general good health.

Exclusion Criteria:

* See above for main selection criteria.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To assess single dose safety and tolerability of an ABT-333 tablet formulation relative to placebo by the evaluation of vital signs, ECGs, physical exams, clinical lab testing and adverse event monitoring | Daily assessment for 5 days then day 30 or more frequently as needed
To evaluate single dose pharmacokinetics of an ABT-333 tablet formulation | Day 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Yamamura, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 19102, Kagoshima, Japan